CLINICAL TRIAL: NCT04790747
Title: Clinical Trial for the Safety and Efficacy of Sequential Radiotherapy With CAR-T Cells in the Treatment of Relapsed and Refractory Hematological Malignancies With Extramedullary Lesions
Brief Title: Sequential Radiotherapy With CAR-T Cells in the Treatment of Relapsed and Refractory Hematological Malignancies With Extramedullary Lesions
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EML-001
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hematological Malignancies
Keywords: radiotherapy; CAR-T; extramedullary lesions; relapsed and refractory
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy and CAR-T therapy (Experimental): sequential radiotherapy and CAR-T cell therapy
  Interventions: Drug: CAR-T cells

INTERVENTIONS:
Drug: CAR-T cells — Each subject receives sequential radiotherapy and CAR-T cells by intravenous infusion

SUMMARY:
Clinical trial for the safety and efficacy of sequential radiotherapy with CAR-T cells in the treatment of relapsed and refractory hematological malignancies with extramedullary lesions

DETAILED DESCRIPTION:
This is a prospective, single arm study. To evaluate the safety and efficacy of sequential radiotherapy with CAR-T cells in the treatment of relapsed and refractory hematological malignancies with extramedullary lesions. The main endpoints were dose limiting toxicity (DLT) and incidence of adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

Age≥15 years old; Relapsed and refractory hematological malignancies with extramedullary lesions, mainly including B-cell non Hodgkin's lymphoma, multiple myeloma, acute lymphoblastic leukemia, etc; Flow cytometry or pathological biopsy confirmed that tumor cells have potential therapeutic targets for Car-T cells; PET-CT confirmed that the extramedullary lesions were located in a single radiotherapy region; Anticipated survival time more than 12 weeks; Those who voluntarily participated in this trial and provided informed consent.

Exclusion Criteria:

History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases; Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past; Pregnant (or lactating) women; Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis); Active infection of hepatitis B virus or hepatitis C virus; Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving inhaled steroids; Previously treated with any CAR-T cell product or other genetically-modified T cell therapies; Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl; Other uncontrolled diseases that were not suitable for this trial; Patients with HIV infection; Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CAR-T cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Complete Remission Rate | up to 28 days after CAR-T cells infusion
  Complete Remission Rate after CAR-T cell therapy
Overall survival (OS) | Up to 2 years after CAR-T cells infusion
  From the first infusion of CD19 CAR-T cells to death or the last visit
Disease-free survival (DFS) | Up to 2 years after CAR-T cells infusion
  From the complete remission to the occurrence of any event, including death, relapse (any one occurs first), and the last visit
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No